CLINICAL TRIAL: NCT07004413
Title: Randomized Study to Compare First-line Treatment With Either Continuous or Intermittent Cetuximab Plus FOLFIRI in Patients With RAS/BRAF-wild-type Metastatic Colorectal Cancer (mCRC): AIO-KRK-0524 / FIRE-11
Brief Title: Continuous or Intermittent Cetuximab Plus FOLFIRI as First-line Treatment in RAS/BRAF Wild-type mCRC Patients
Acronym: FIRE-11
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Merck Healthcare Germany GmbH, an affiliate of Merck KGaA, Darmstadt, Germany (Unknown); Guardant Health, Inc. (Industry)
Responsible Party: Principal Investigator, Sebastian Stintzing, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1319-8357; 2025-522377-12-00 (EU CTIS Number); AIO-KRK-0524 (Other: German working group for medical oncology (Arbeitsgemeinschaft Internistische Onkologie (AIO)))
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Metastatic colorectal cancer; RAS; BRAF; cetuximab; ctDNA; treatment break
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: open-label, randomized, controlled, multicenter, phase III study with two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFIRI+cetuximab, continuously applied (Active Comparator): Continuous application of FOLFIRI+cetuximab until disease progression according to standard of care
  Interventions: Drug: FOLFIRI+cetuximab
- FOLFIRI+cetuximab, applied with scheduled treatment breaks (Experimental): Scheduled treatment break after up to 6 cycles of FOLFIRI+cetuximab until radiological (or, in part 2, ctDNA-based) disease progression
  Interventions: Drug: FOLFIRI+cetuximab; Diagnostic Test: Guardant360 ctDNA assay

INTERVENTIONS:
Drug: FOLFIRI+cetuximab — Cetuximab 500 mg/m², 90 min IV infusion on d1; Irinotecan: 180 mg/m², 90-120 min IV infusion on d1; Folinic acid: 400mg/m², 1-2h IV Infusion on d1; 5-FU: 2400 mg/m², 46 h IV infusion on d1. Cycles are repeated on day 15.
  Other Names: Cetuximab, Irinotecan, Folinic acid, 5-fluorouracil (FU)
Diagnostic Test: Guardant360 ctDNA assay — Determination of circulating tumor DNA (ctDNA) in the peripheral blood, part 1: retrospective threshold determination to predict radiological disease progression in Arm 2; part 2: prospective validation of the in part 1 identified ctDNA threshold to guide the scheduled treatment breaks and treatment in Arm 2
  Arms: FOLFIRI+cetuximab, applied with scheduled treatment breaks

SUMMARY:
The goal of this clinical trial is to learn if the application of the chemotherapy FOLFIRI and cetuximab works better when given with scheduled breaks or continuously in adults with metastatic colorectal cancer. The main question it aims to answer is, whether worsening of disease after 12 months of treatment is lower when the treatment is given with breaks or given continuously. It will also answer the question whether the quality of life is better and side effects are less if chemotherapy is given with breaks.

Additionally, the treatment breaks will be controlled by blood tests and imaging examinations. A novel blood test will be introduced to investigate, whether worsening of the disease might be detected before the imaging, and whether a quicker reaction by re-starting the therapy would help the patients.

Participants will:

* receive an established chemotherapy mit FOLFIRI and cetuximab
* Receive blood tests every 4 weeks and imaging investigations every 12 weeks
* fill out questionnaires to report their quality of life

DETAILED DESCRIPTION:
This is a combined multicenter, randomized phase III clinical trial and interventional clinical performance study according to IVDR investigating the superiority of intermittent application of FOLFIRI plus cetuximab followed by a scheduled treatment pause compared to continuous treatment with FOLFIRI plus cetuximab until disease progression or unacceptable toxicity. This study is accompanied by a translational research program.

This study protocol is driven by a CTR-conform question and primary endpoint, the PFS from randomization to progression on treatment at 12 months, and supplemented by a separate, complementary, interventional clinical performance study to assess ctDNA as biomarker of early disease progression as a key secondary endpoint. Details regarding the IVD part are specified in the complementary interventional clinical performance study protocol.

Treatment is planned until progression, death or unacceptable toxicity. Patients are followed up with regard to survival and if applicable subsequent anti - cancer treatments until death or -after end of study treatment- for at least 3 years after start of treatment, whichever date is earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's signed informed consent
2. Histologically confirmed, UICC stage IV unresectable adenocarcinoma of the colon or rectum
3. Locally confirmed RAS/BRAF wild-type tumor status (KRAS and NRAS exon 2, 3, 4, BRAF exon 11/15)

   a) Note: A maximum of two cycles FOLFIRI is allowed prior to start of induction treatment until the molecular characterization is fully reported
4. Centrally confirmed RAS/BRAF wild-type status by liquid biopsy during screening phase
5. Age 18 or older at the time of written informed consent
6. ECOG performance status below or equal 1
7. Presence of at least one measurable reference lesion according to the RECIST 1.1 criteria
8. Archival tumor tissue available
9. Consent to storage, molecular and genetic profiling of tumor material and blood
10. Adequate bone marrow function:

    1. Leukocytes ≥ 3.0 x 109/L with neutrophils ≥ 1.5 x 109/L
    2. Thrombocytes ≥ 100 x 109/L
    3. Hemoglobin ≥ 8 g/dL)
11. Adequate hepatic function:

    1. Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
    2. ALAT and ASAT ≤ 2.5 x ULN (in the presence of hepatic metastases, ALAT and ASAT ≤ 5 x ULN)
    3. INR < 1.5 and aPTT < 1.5 x ULN (patients without anticoagulation). Therapeutic anticoagulation is allowed if INR and aPTT have remained stable within the therapeutic range for at least 2 weeks.
12. Adequate renal function:

    a) Creatinine clearance (calculated according to Cockcroft and Gault) ≥ 50 mL/min
13. Proficient fluorouracil metabolism as defined:

    1. Prior treatment with 5-FU or capecitabine without unusual toxicity OR
    2. If tested, normal DPD deficiency test according to the standard of the study site OR
    3. If tested, in patients with DPD deficiency test with a CPIC activity score of 1.0-1.5 fluoropyrimidine dosage should be reduced by 50%
14. Females of childbearing potential (FCBPs) and men must agree to use highly effective contraceptive measures (Pearl index <1) or practice true abstinence from any heterosexual intercourse (true abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject) for the duration of the study treatment and for at least 6 months after last administration of study medication. A woman will be considered as being of childbearing potential unless she is at least 50 years old and moreover has gone through menopause for at least 2 years or has been surgically sterilized. For men: With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 6 months after the last dose of study treatment. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 6 months after the last dose of study medication to avoid exposing the embryo.

Exclusion Criteria:

1. Proof of a RAS or BRAF mutation (KRAS/NRAS exons 2, 3, 4 or BRAF exon 15) in the tumor (proven in the primary tumor or metastasis) or liquid biopsy during screening phase.
2. Previous chemotherapy for the colorectal cancer with the exception of adjuvant treatment, completed at least 6 months before written informed consent.
3. New York Heart Association Class III or greater heart failure by clinical judgement.
4. Myocardial infarction, balloon angioplasty (PTCA) with or without stenting, and cerebral vascular accident/stroke within the past 12 months before randomization
5. Unstable angina pectoris
6. Unstable cardiac arrhythmia > grade 2 NCI CTCAE despite anti-arrhythmic therapy.
7. Active uncontrolled infection by investigator's perspective.
8. Pre-existing pulmonary fibrosis or immune pneumonitis
9. Additional cancer treatment (chemotherapy, radiation, immunotherapy or hormone treatment) during the study treatment in first-line and third-line treatment (treatments that are conducted as part of an anthroposophical or homeopathic treatment approach, e.g. mistletoe therapy does not represent an exclusion criterion)
10. Participation in a clinical study or experimental drug treatment within 30 days prior to written informed consent or within a period of 5 half-lives of the substances administered in a clinical study or during an experimental drug treatment prior to written informed consent, depending on which period is longest or simultaneous participation in another study while taking part in the study
11. Known hypersensitivity or allergic reaction to any of the following substances: 5-fluorouracil, folinic acid, cetuximab, irinotecan and chemically related substances and/or hypersensitivity to any of the components in the formulations of the aforementioned substances, including known hypersensitivity reactions to monoclonal antibodies NCI CTC grade ≥ 3.
12. Known hypersensitivity to Chinese hamster ovary cell (CHO) -cellular products or other recombinant human or humanized monoclonal antibodies
13. Patients with known brain metastases or leptomeningeal disease. In case of clinical suspicion of brain metastasis, a cranial CT or MRI must be performed to rule out brain metastasis before study inclusion.
14. History of acute or subacute intestinal occlusion, inflammatory bowel disease, immune colitis or chronic diarrhea
15. Symptomatic peritoneal carcinosis
16. Severe, non-healing wounds, ulcers or bone fractures
17. Requirement for immunization with live vaccine including attenuated live vaccine from at least 4 weeks before begin of induction treatment until 6 months after the administration of IMPs.
18. Hemorrhagic diathesis or known thrombophilia
19. Known glucuronidation deficiency (Gilbert's syndrome) (specific screening not required)
20. Treatment with nucleoside analogues including sorivudine or brivudine within 28 days before begin of induction treatment or requirement for concomitant antiviral treatment with sorivudine or brivudine or analogues
21. History of a second primary malignancy during the past 5 years before written informed consent or during participation in the study, with the exception of a basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ, if these were treated curatively.
22. Active alcohol or drug abuse
23. Any significant adverse event that has not adequately resolved, severe acute or chronic concomitant disease or medical condition including psychiatric conditions (including recent i.e. within the past year or active suicidal ideation or behavior) or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
24. Absent or restricted legal capacity
25. Patients who are institutionalized by order of court or public authority
26. Patients who might be dependent on the sponsor/investigator or the trial site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) on treatment rate at 12 months | 12 months
  Percentage of patients who did not experience disease progression or death, whichever occurs first, while receiving active treatment for 12 months starting from randomization.

SECONDARY OUTCOMES:
PFS1 to PFSN | up to 24 months
  Each PFS from treatment start with FOLFIRI+cetuximab to the first disease progression in the respective treatment period
Overall survival (OS) | At least 5 years after randomization
  Time from randomization to the date of death by any cause
Objective Response Rate (ORR) | up to 24 months
  Radiological objective response as determined by RECIST 1.1 criteria
Dynamics of the tumor markers CEA and CA19-9 | Up to 24 months
Early Tumor Shrinkage (ETS) | 8 weeks
  Radiological reduction of tumor volume by 20% at the first re-staging (8 weeks)
Depth of Response (DpR) | up to 24 months
  Maximum relative decrease of radiologically determined tumor mass in percent
Circulating tumor DNA (ctDNA) as additional prospective biomarker of serum RAS/BRAF wild-type status and predictor early radiological disease progression | Up to 24 months
  Prospective validation to use ctDNA based RAS/BRAF mutational analysis in addition to tissue-based RAS/BRAF testing to exclude RAS/BRAF mutant tumors from treatment, definition and validation of a threshold value in ctDNA change predicting progressive disease during treatment pause
Quality of Life (QoL) | up to 24 months
  QoL as assessed with the QoL questionnaire EQ-5D-5L
Adverse events | up to 24 months
  Type, incidence, severity, and causal relationship to IMPs of non-serious adverse events and serious adverse events (severity evaluated according to CTCAE version 5.0)

OTHER OUTCOMES:
Translational research | up to 5 years
  DNA, mRNA and protein expression derived from FFPE tumor tissue and longitudinal blood samples, role of molecular hyperselection on treatment efficacy, integration of digital pathology using digitalized stained tumor tissue sections

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No